CLINICAL TRIAL: NCT06666426
Title: A Randomized, Controlled Trial on the Safety, Efficacy, and Patient Reported Experience Comparing PureWick™ System With an Established Comparator Overnight in the Home Setting (PUREST)
Brief Title: This Study Will Collect Clinical and Patient Reported Experience Data From Participants Requiring Urine Output Management Overnight in the Home Setting.
Acronym: PUREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCC-23HC009
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Adult Nocturnal Enuresis; Urinary Incontinence (UI)
Keywords: nighttime urinary incontinence; Quality of Life; sleep disturbance; NQoL; PROMIS; Purewick; Hollister; females; PureWick Flex Female External Catheter; PureWick Urine Collection System; The Hollister Female Urinary Pouch; BD; Becton, Dickinson and Company
MeSH Terms: conditions — Nocturnal Enuresis; Urinary Incontinence; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hollister (Active Comparator)
  Interventions: Device: Hollister Female Urinary Pouch External Collection Device
- PureWick (Experimental)
  Interventions: Device: PureWick System

INTERVENTIONS:
Device: PureWick System — The PureWick System consists of the PureWick Urine Collection System used with the PureWick Flex Female External Catheter, which are intended for non-invasive urine output management.
  Arms: PureWick
Device: Hollister Female Urinary Pouch External Collection Device — The Hollister Female Urinary Pouch External Collection Device is intended to collect and contain urine for individuals with urinary incontinence.
  Arms: Hollister

SUMMARY:
This post-market study will assess the performance of and user experience with the PureWick™ System in a home setting. The study will also observe safety of the study device and collect information from participants about their quality of life before and after using the device.

DETAILED DESCRIPTION:
Approximately 150 women with nighttime urinary incontinence will take part in this prospective, open-label, randomized trial. Participants will use one of two different study devices during the study to manage urine output at night: PureWick™ System or the Hollister® Female Urinary Pouch External Collection Device. Participant device assignment will be random. Participants will use the assigned urine management device overnight while sleeping and will be followed for approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female Participants greater than or equal to 18 years of age at the time of signing the informed consent.
2. Currently use diapers or equivalent at night for urine output management.
3. Willing to comply with all study procedures in this CIP.
4. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Has frequent episodes of bowel incontinence without a fecal management system in place; or
2. Has moderate to heavy menstruation and cannot use a tampon or menstrual cup; or
3. Has urinary tract, vaginal or other chronic infections, active genital herpes; or
4. Has urinary retention; or
5. Is agitated, combative, and/or uncooperative and may remove the external catheter or pouch; or
6. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
7. Has any pre-existing neurological, psychiatric, or other condition that would confound quality of life assessment or would make it difficult to self-report on quality-of-life questionnaires in the opinion of the investigator; or
8. Is known to be pregnant at time of enrollment (for women of childbearing age); or
9. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Performance of the PureWick System in the home setting | From enrollment to the end of treatment at 4 weeks
  Daily capture rate (captured as % of urine captured by device and collected in canister, measured by weight)
Safety of the PureWick System in the home setting | From enrollment to the end of treatment at 4 weeks
  Daily skin irritation score using the 5-point Draize dermal irritation scoring system ranging from 0 to 4 with higher scores indicating greater irritation.

SECONDARY OUTCOMES:
Participant Device Tolerance | From enrollment to the end of treatment at 4 weeks
  Number of days of actual device use over the expected treatment duration.
Participant Device Experience - Comfort | From enrollment to the end of treatment at 4 weeks
  Overall comfort on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome.
Participant Device Experience - Ease of Use | From enrollment to the end of treatment at 4 weeks
  Overall ease of use on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome.

OTHER OUTCOMES:
Nocturnal Incontinence related Quality of Life | From enrollment to the end of treatment at 4 weeks
  Nocturia Quality of Life (N-QOL) score collected at baseline and every 2 weeks during treatment with higher scores indicating better QoL. The NQoL contains 12 scored items each scored from 0 to 4. All item scores are computed into a total score ranging from 0-100 where 0 is the worst QoL and 100 is the best QoL.
Participant Sleep Quality | From enrollment to the end of treatment at 4 weeks
  PROMIS Sleep Disturbance Short Form 4a score collected at baseline and every 7 days during treatment with higher scores indicating greater sleep disturbance.
  The PROMIS Sleep Disturbance 4a contains 4 scored items each scored from 1 to 5. All item raw scores are computed into a total score where higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Lakeview Clinical Research, Guntersville, Alabama
  - New Horizons Clinical Trials, Chandler, Arizona
  - The Practice of Medicine INC., Eagle Rock, California
  - Finlay Medical Research, Greenacres City, Florida
  - Finlay Medical Research, Miami, Florida
  - Smith Medical Center, Dunwoody, Georgia
  - Sonar Clinical Research, Riverdale, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Research Integrity, Owensboro, Kentucky
  - Revive Research Institute, Dearborn Heights, Michigan
  - Trialfinity Clinical Research Center, Hamilton, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Prime Global Research, The Bronx, New York
  - MultiSpecialty Clinical Research, Johnson City, Tennessee
  - Trio Clinical Trials, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medina JC, Fakih M, Khalsa S, Redmond D, Kennelly MJ. Safety, Efficacy, and Patient-Reported Outcomes of the PureWick System Versus Comparator for Nocturnal Urinary Incontinence in the Home Setting: Results of a Randomized Trial. J Clin Med. 2025 Dec 9;14(24):8699. doi: 10.3390/jcm14248699. PMID 41464602